CLINICAL TRIAL: NCT04066803
Title: Safety and Efficacy of Optimal Methotrexate With Folic Acid in Patients With Rheumatoid Arthritis in Meizhou, Guangdong: a Randomized Case-control Study
Brief Title: Optimal MTX Dose With Folic Acid Randomized Case-control Trial
Acronym: MTXFARCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Principal Investigator, Gu Jieruo, Rheumatology Department, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QHJH201805
Record Dates: First submitted 2018-12-11; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid; Antirheumatic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTX group with folic acid (Experimental): the group with optimal MTX dose (gradually increased from 0 to 12weeks，appropriate folic acid，and stable original other DMARDs
  Interventions: Drug: MTX; Drug: Folic Acid; Drug: DMARDs
- control group without folic acid (Active Comparator): the group with stable MTX 10mg/w dose and maximum DMARDs doses（graduallly increased from 0 to 12 weeks）without folic acid
  Interventions: Drug: MTX; Drug: DMARDs

INTERVENTIONS:
Drug: MTX — MTX group would be intervened by incremental MTX and folic acid，while the control group would be intervened by incremental original DMARDs they already used（including Leflunomide，Hydroxychloroquine,Sulfasalazine,Azathioprine,Tripterygium glycosides and Total glucosides of paeony)
Drug: Folic Acid — MTX group would be intervened by folic acid，while the control group would be not intervened by folic acid
  Arms: MTX group with folic acid
Drug: DMARDs — including Leflunomide，Hydroxychloroquine,Sulfasalazine,Azathioprine,Tripterygium glycosides and Total glucosides of paeony

SUMMARY:
This is an open, single-center, randomized,case controlled, prospective study. Previous studies in China lacked data of efficacy and safety of optimal methotrexate (MTX) dose with/without other anti-rheumatoid drugs (DMARDs) in the treatment of rheumatoid arthritis (RA) .Meanwhile there was no study on the optimal folic acid dose in aspect of preventing side effects of MTX. So we designed the experiment below.

The research planned to recruit 160 RA patients in Meizhou, Guangdong Province,China. The volunteers had no relief with 10 mg of MTX per week with/without other DMARDs for at least 3 month. They were randomly divided into 1:1 groups. The experimental group would be treated with original dMARDs ,incremental MTX( gradually increased to the optimal dose (0.3 mg/kg) in the first 12 weeks）and folic acid (the dose adjusted as appropriate with range from 5 mg to 90 mg per week) . While the control group would be treated with original MTX（10mg per week) and incremental original dMARDs( gradually increased to the maximum dose in the first 12 weeks). The two groups would keep the 12th week treatment last to the 36th week, and the efficacy and safety indexes would be evaluated during the whole study.

The objective of the study was to determine the efficacy and safety of the optimal dose of MTX in Chinese patients with rheumatoid arthritis, and to determine the efficacy and optimal prevention dose of folic acid in Chinese RA patients. It might be helpful for Chinese rheumatologists to use MTX accurately and efficiently to treat RA patients in clinical work.

ELIGIBILITY:
Inclusion Criteria:

1. According to the revised 1987 American Academy of Rheumatology (ACR) RA classification criteria, subjects must be diagnosed as rheumatoid arthritis ≥6 months.
2. MTX was given 10 mg/week（not the maximum dose of MTX (calculated as 0.3 mg/kg)) for ≥3 months before admission.
3. At the screening and baseline phases, the number of swollen joints (SJC) should be ≥1 (counting 66 joints), and the number of tender joints (TJC) should be ≥ 1 (counting 66 joints); the ESR should be ≥20 mm/h, and/or the CRP should be ≥ 10 mg/l;
4. The age of the subjects ranged from 18 to 70 years.
5. The following RA drugs can be used in combination within 3 months before admission; oral glucocorticoid (prednisone ≤10 mg/d or its equivalent), non-steroidal anti-inflammatory drugs (≤ the maximum recommended dose), leflunomide, hydroxychloroquine, sulfasalazine, total paeoniflorin, Tripterygium glycoside, azathioprine, and MTX. The stable dose of DMARDs should be at least 4 weeks before baseline, and the combined dose of DMARDs beside MTX could not reach the full dose.
6. Women of childbearing age should agree to take effective contraceptive measures during the trial period;
7. The urinary pregnancy test of women of childbearing age was negative at screening time.
8. Understand the steps and contents of the experiment and sign the informed consent to participate in the experiment.

Exclusion Criteria:

1. Those who underwent major surgery (including joint surgery) within 8 weeks before screening or who planned major surgery within 6 months after random selection;
2. Patients with autoimmune diseases except RA include SLE, MCTD, scleroderma and polymyositis. But subjects with RA and secondary Sjogren syndrome were allowed to participate in the trial.
3. Inflammatory arthritis (such as gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) .
4. Intra-articular injection or other injection of corticosteroids within 4 weeks before baseline;
5. Those who had been vaccinated with live/inactivated vaccine within 4 weeks before baseline;
6. Three months before admission, the following drugs were used: cyclophosphamide, biological agents and folic acid.
7. DMARDs dose reached maximum dosage in 3 months before admission， or DMARDs≥3 were used in 3 months before admission
8. Subjects with severe uncontrolled diseases including cardiovascular disease, nervous system disease, pulmonary disease (including obstructive pulmonary disease and interstitial lung disease), nephropathy, liver disease, endocrine disease (including uncontrolled diabetes mellitus) and gastrointestinal diseases;
9. known history of active or recurrent bacterial, viral, fungal, Mycobacterium or other infections (including, but not limited to, tuberculosis and atypical mycobacterium diseases, chest X-rays showing granulomatous diseases, hepatitis B and C, HIV infection, herpes zoster, but excluding Onychomycosis) ，any infection requiring hospitalization and intravenous antibiotic therapy within 4 weeks before screening ，or oral antibiotic therapy within 2 weeks before screening; active hepatitis B refers to HBsAg-positive patients without antiviral drugs and HBV-DNA > 10^4; active hepatitis C refers to anti-HCV-positive patients without antiviral drugs and HCV-RNA > 10^4;
10. Subjects with a history of malignant tumors, including solid tumors and hematological malignancies (except excised or cured skin basal cell carcinomas);
11. Pregnant or lactating women (breastfeeding);
12. Subjects with neuropathy and other painful diseases may interfere with pain assessment.
13. Serum creatinine > 1.5 mg/dl (equivalent to 133 umol/L);
14. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times of the upper limit of normal value (if ALT or AST is greater than 2 times of the upper limit of normal value for the first time, it should be sampled again during the screening period), or total bilirubin is greater than the upper limit of normal value (if total bilirubin is greater than the upper limit of normal value for the first time at the screening, sampling should be done again during the selection period).
15. Platelet count < 100 x 10^9/L, or white blood cells < 3 x 10^9/L;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
The response rate of ACR20 at the 36th weeks | at the 36th weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yun Feng Pan, Master, Study Director — the 3rd Hospital of Sun Yat-sen University
Locations (1):
- the 3rd Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
No plan to share.

REFERENCES:
- [Result] Gaujoux-Viala C, Rincheval N, Dougados M, Combe B, Fautrel B. Optimal methotrexate dose is associated with better clinical outcomes than non-optimal dose in daily practice: results from the ESPOIR early arthritis cohort. Ann Rheum Dis. 2017 Dec;76(12):2054-2060. doi: 10.1136/annrheumdis-2017-211268. Epub 2017 Sep 2. PMID 28866645